CLINICAL TRIAL: NCT04817423
Title: Automated ICD Coding of Primary Diagnosis Based on Machine Learning
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-1425
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Model training and test group: Data set will be split into training group and test group, where training group will be used for model building, and test group for subsequent evaluation and verification.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study aims to develop and validate machine learning model in ICD-10 coding of primary diagnosis related to cardiovascular diseases in Chinese corpus.

DETAILED DESCRIPTION:
The accuracy and productivity of ICD coding has always been a concern of clinical practice. Errors of ICD codes may result in claim denials and missed revenue. However, ICD coding process is complex, time-consuming and error-prone. More experienced coders are in need, but there is an increasing lack of supply. Automated ICD coding has potential to facilitate clinical coders for improved efficiency and quality. Model performance of related studies is still far below coders and both the accuracy and interpretability need to be improved in great demand. Besides, studies in Chinese corpus are not sufficient.

In this study, the investigators will implement automated ICD coding study based on inpatient' data collected from electronic medical records from Fuwai Hospital, the world's largest medical center for cardiovascular disease. Feature engineering and machine learning methods will be used to develop classification models with good performance, interpretability and practicability for ICD codes of primary diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Admissions in Fuwai Hospital, from January 1, 2019, to December 31, 2020

Exclusion Criteria:

* Admissions stayed in nephrology department, Fuwai Hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Admissions in Fuwai Hospital
Sampling Method: Non-Probability Sample
Enrollment: 74880 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
ICD code of primary diagnosis | At the end of enrollment
  Each admission will be a sample in this study. The ICD code of primary diagnosis assigned by medical coders for each admission will be collected as the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, PhD, Principal Investigator — China National Center for Cardiovascular Diseases
Locations (1):
- Fuwai Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No